CLINICAL TRIAL: NCT00938821
Title: The Use of Very Low Dose Caudal Morphine for Postoperative Pain Management in Out Patients
Brief Title: Very Low Dose Caudal Morphine for Postoperative Pain Management
Status: Completed | Type: Observational
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Other Study IDs: 15028
Record Dates: First submitted 2009-07-09; First posted 2009-07-14 (Estimated); Last update posted 2017-11-21 (Actual); Status verified 2017-11

CONDITIONS: Caudal Anesthesia
MeSH Terms: interventions — Morphine; Bupivacaine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Caudal Block: Review of charts of patients that received very low dose morphine administered caudally (M) and plain caudal block with Ropivacaine or Marcaine (B).
  Interventions: Procedure: Caudal block

INTERVENTIONS:
Procedure: Caudal block — Chart review of patients that received very low dose morphine administered caudally (M) and plain caudal block with Ropivacaine or Marcaine (B)from October 2008 to October 2009.
  Other Names: Postoperative pain; Morphine; Bupivacaine

SUMMARY:
This is a chart review. The aim of this study is to investigate the effectiveness and side effects of very low dose morphine administered caudally to children that went to surgical procedures that used caudal anesthesia. The study compares caudal block with Bupivacaine (1 ml kg_1 of bupivacaine 0.25% and saline 0.02 ml kg_10) with very low dose morphine (a mix of 1 ml kg_-1 of ropivacaine 0.2% and preservative-free morphine: 10 µg kg-1).

DETAILED DESCRIPTION:
Caudal anesthesia is the most common technique of epidural anesthesia in children. Caudal anesthesia is recommended for most surgical procedures of the lower part of the body, including herniorrhaphies; operations on the urinary tract, anus, and rectum; and orthopedic procedures on the pelvic girdle and lower extremities. Many anesthetic agents have been used for caudal anesthesia in pediatric patients, with lidocaine and Bupivacaine being most common. The major problems associated with this technique are the limited duration of analgesia and unwanted motor blockade.

Addition of medications that prolong analgesia after a single shot caudal block has been investigated. Several authors have mentioned a special interest in using an opioid like morphine in caudal block for postoperative analgesia. When low dose morphine is used, the side effects are lower than when higher dose of morphine are used. A larger and definitive study is needed to compare very low dose morphine via caudal administration and caudal block without Opioid with regard to duration of analgesia and frequency of side effects. We plan to conduct a chart review in our center on pediatric patients that went to urological, orthopedic, and general surgery procedures for which caudal block were given and compare the effectiveness and side effects of very low dose morphine and caudal block without Opioid.

ELIGIBILITY:
Inclusion Criteria:

* The subject did have elective Urological procedures such us circumcision, orchidopexy and inguinal hernia repair, orthopedic and general surgery procedures for which caudal block are usually administered for pain management.

Exclusion Criteria:

* Subjects with non elective or emergency surgery (must have the surgery no matter what).
* Subjects with surgical procedures that are not planned to be conducted with the use of general anesthesia. Subjects that are not allowed to receive the anesthesia agents indicated per protocol and general anesthesia.
* American Society of Anesthesiologists, Physical Status classification greater than 2 (uncontrolled systemic disease or more than one systemic disease).
* Patients with a history of chronic pain conditions.
* Infection around the sacral hiatus.
* Coagulopathy.
* Anatomic abnormalities.
* Patient with mentally retardation.
* Patient with history of attention deficit and/or behavioral problems.

Ages: 1 Month to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: This is a chart review from October 2008 to October 2009 of children from 1 month of age to 10 years old that went to elective Urological procedures such us circumcision, orchidopexy and inguinal hernia repair, orthopedic and general surgery procedures for which caudal block are usually administered for pain management
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2010-01; Primary Completion 2012-12-11 (Actual); Study Completion 2012-12-11 (Actual)

PRIMARY OUTCOMES:
The study's primary research question, which relates to between-group differences is duration of analgesia. | 1 year 5 months

SECONDARY OUTCOMES:
Between-group differences in the proportion of patients clinically significant side effects will be assessed. | 1 year 5 months

CONTACTS AND LOCATIONS:
Overall Officials: Alberto J. de Armendi, MD, AM, MBA, Principal Investigator — Oklahoma University Health Sciences Center
Locations (1):
- The University of Oklahoma Health Sciences Center Deparment of Anesthesiology, Oklahoma City, Oklahoma, United States

REFERENCES:
- [Background] Tsui BC, Berde CB. Caudal analgesia and anesthesia techniques in children. Curr Opin Anaesthesiol. 2005 Jun;18(3):283-8. doi: 10.1097/01.aco.0000169236.91185.5b. PMID 16534352
- [Background] Mayhew JF, Brodsky RC, Blakey D, Petersen W. Low-dose caudal morphine for postoperative analgesia in infants and children: a report of 500 cases. J Clin Anesth. 1995 Dec;7(8):640-2. doi: 10.1016/0952-8180(95)00089-5. PMID 8747562
- [Background] Krane EJ, Tyler DC, Jacobson LE. The dose response of caudal morphine in children. Anesthesiology. 1989 Jul;71(1):48-52. doi: 10.1097/00000542-198907000-00009. PMID 2751139
- [Background] Kawaraguchi Y, Otomo T, Ota C, Uchida N, Taniguchi A, Inoue S. A prospective, double-blind, randomized trial of caudal block using ropivacaine 0.2% with or without fentanyl 1 microg kg-1 in children. Br J Anaesth. 2006 Dec;97(6):858-61. doi: 10.1093/bja/ael249. Epub 2006 Sep 13. PMID 16973647
- [Background] Cyna AM, Middleton P. Caudal epidural block versus other methods of postoperative pain relief for circumcision in boys. Cochrane Database Syst Rev. 2008 Oct 8;2008(4):CD003005. doi: 10.1002/14651858.CD003005.pub2. PMID 18843636
- [Background] Hong D, Flood P, Diaz G. The side effects of morphine and hydromorphone patient-controlled analgesia. Anesth Analg. 2008 Oct;107(4):1384-9. doi: 10.1213/ane.0b013e3181823efb. PMID 18806056
- [Background] Eschertzhuber S, Hohlrieder M, Keller C, Oswald E, Kuehbacher G, Innerhofer P. Comparison of high- and low-dose intrathecal morphine for spinal fusion in children. Br J Anaesth. 2008 Apr;100(4):538-43. doi: 10.1093/bja/aen025. Epub 2008 Feb 27. PMID 18305080
- [Background] Castillo-Zamora C, Castillo-Peralta LA, Nava-Ocampo AA. Dose minimization study of single-dose epidural morphine in patients undergoing hip surgery under regional anesthesia with bupivacaine. Paediatr Anaesth. 2005 Jan;15(1):29-36. doi: 10.1111/j.1460-9592.2004.01391.x. PMID 15649160
- [Background] Tyler DC, Krane EJ. Epidural opioids in children. J Pediatr Surg. 1989 May;24(5):469-73. doi: 10.1016/s0022-3468(89)80404-x. PMID 2567780
- [Background] Cesur M, Alici HA, Erdem AF, Yapanoglu T, Silbir F. Effects of reduction of the caudal morphine dose in paediatric circumcision on quality of postoperative analgesia and morphine-related side-effects. Anaesth Intensive Care. 2007 Oct;35(5):743-7. doi: 10.1177/0310057X0703500514. PMID 17933162
- [Background] Mayhew J, Siddiqui S. Very low dose of caudal morphine. Paediatr Anaesth. 2005 Jul;15(7):623. doi: 10.1111/j.1460-9592.2005.01662.x. No abstract available. PMID 15960653
- [Background] Voepel-Lewis T, Merkel S, Tait AR, Trzcinka A, Malviya S. The reliability and validity of the Face, Legs, Activity, Cry, Consolability observational tool as a measure of pain in children with cognitive impairment. Anesth Analg. 2002 Nov;95(5):1224-9, table of contents. doi: 10.1097/00000539-200211000-00020. PMID 12401598